CLINICAL TRIAL: NCT00082342
Title: Transcranial Direct Current Stimulation for the Treatment of Parkinson's Disease
Brief Title: Transcranial Direct Current Stimulation to Treat Symptoms of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Mark Hallett, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 030116; 03-N-0116
Record Dates: First submitted 2004-05-06; First posted 2004-05-06 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson Disease
Keywords: Human Brain; Electrical Stimulation; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- real transcranial direct current stimulation (tDCS) (Active Comparator)
  Interventions: Device: Phoressor II (IOMED)
- sham transcranial direct current stimulation (tDCS) (Sham Comparator)
  Interventions: Device: Phoressor II (IOMED)

INTERVENTIONS:
Device: Phoressor II (IOMED) — sham stimulation
  Arms: sham transcranial direct current stimulation (tDCS)
Device: Phoressor II (IOMED) — real tDCS stimulation
  Arms: real transcranial direct current stimulation (tDCS)

SUMMARY:
This study will examine the effects of transcranial direct current stimulation (tDCS) on gait (walking) problems and rigidity in patients with Parkinson's disease. tDCS is a method of brain stimulation that may be able to change the electrical activity of the nerves of the brain, possibly causing Parkinson's disease symptoms to improve.

Patients between 40 and 80 years of age with moderately severe Parkinson's disease whose main symptoms are problems with walking, including freezing, or rigidity, may be eligible for this study. Candidates must be taking Sinemet or another L-DOPA drug and not have too much tremor.

Participants will be assigned to receive either real or sham (placebo) tDCS. Both groups will have eight treatments over 3-1/2 weeks. For the tDCS, electrodes are placed on wet pads on the scalp. An electrical current passes through the electrodes, travels through the scalp and skull, and causes small electrical currents in the cortex-the outer part of the brain. Participants will have a neurological examination, including an evaluation of walking, just before and just after each tDCS session. Patients' motor function will be re-evaluated at 1, 3, and 6 months after the last tDCS treatment.

...

DETAILED DESCRIPTION:
The treatment of Parkinson's disease (PD) needs further improvement, particularly in the areas of gait and freezing. Transcranial direct current stimulation (tDCS) which passes weak direct current (DC) current through the skull and across the cortex has been done for many years with numerous effects described in healthy subjects and patients with mental illness. Recently, it has been shown by objective means, in controlled experiments, that this type of treatment has robust and lasting effects on the excitability of the motor cortex in healthy humans. We hypothesize that tDCS will have a beneficial effect on gait and freezing in medicated patients, and we propose to test this in a controlled trial. Specifically, we propose to look at the effect of 1-2 mA tDCS with anode position over the frontal poles and/or premotor and primary motor cortex, and cathode over mastoid process. Over a one-year period, we will enroll 42 adults with PD and evaluate the acute tDCS effects over a period of four weeks (eight tDCS sessions, nine visits). Additional ratings will be done at one and three months after the end of tDCS sessions. Symptoms will be evaluated with standard tests of motor function, including the Unified Parkinson's Disease Rating Scale (UPDRS) and specific tests of gait and freezing. We will also look for cumulative, long-lasting effects over the three-month period.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with PD corresponding to inclusion criteria will be recruited from the Human Motor Control Section Clinic (HMCS).

Subjects will be men and women aged 40-80 years with DOPA-responsive, akinetic-rigid PD.

Patients who have never participated in HMCS protocols for PD will be interviewed and examined by either the principal investigator or a physician from the Brain Stimulation Unit or HMCS in order to establish the diagnosis of PD and rule out any neurological condition. Only patients with a Hoehm and Yahr grade of 2 to 4 while "off" will be accepted.

Patients must be on a regimen including levodopa. The total dose of levodopa and dopamine agonists (using dopamine equivalents) has to be equal to or more than 375 milligrams per day. Other anti-parkinsonian medications are also acceptable.

Patients should have problems with walking, including freezing, so that their gait time for a 10-meter distance will be six seconds or more.

EXCLUSION CRITERIA:

Exclusion criteria are any significant medical or psychiatric illnesses (except those symptoms often associated with PD or levodopa therapy, such as sundowning and benign hallucination), pallidotomy, implanted electrodes and generator for deep brain stimulation, pregnancy.

Persons with surgically or traumatically implanted foreign bodies such as a pacemaker, implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during TEP will also be excluded. Most of these exclusions also come under the category of significant medical illness.

Patients for whom participation in the study would, in the opinion of the investigators, cause undue risk or stress for reasons such as tendency to fall, excessive fatigue, general frailty, or excessive apprehensiveness will also be excluded.

Patients unable to walk a 10-meter distance will be excluded.

Mentally impaired patients having no capacity to provide their own consent will be excluded from the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-03; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agnew WF, McCreery DB. Considerations for safety in the use of extracranial stimulation for motor evoked potentials. Neurosurgery. 1987 Jan;20(1):143-7. doi: 10.1097/00006123-198701000-00030. PMID 3808255
- [Background] Antal A, Nitsche MA, Paulus W. External modulation of visual perception in humans. Neuroreport. 2001 Nov 16;12(16):3553-5. doi: 10.1097/00001756-200111160-00036. PMID 11733710
- [Background] Braun BL. Treatment of an acute anterior disk displacement in the temporomandibular joint. A case report. Phys Ther. 1987 Aug;67(8):1234-6. doi: 10.1093/ptj/67.8.1234. PMID 3615594
- [Derived] Benninger DH, Lomarev M, Lopez G, Wassermann EM, Li X, Considine E, Hallett M. Transcranial direct current stimulation for the treatment of Parkinson's disease. J Neurol Neurosurg Psychiatry. 2010 Oct;81(10):1105-11. doi: 10.1136/jnnp.2009.202556. PMID 20870863

RESULTS

PARTICIPANT FLOW:
Groups:
- Real tDCS: Transcranial direct current stimulation (tDCS) is a method of non-invasive brain stimulation whereby a direct current is applied to the brain via surface electrodes on the head for a specified time period. It is a form of neurostimulation. Subjects receiving real transcranial direct current stimulation underwent 8 sessions during a 2 1/2 week period while "on" medication. A battery driven stimulator, Phoresor II Model PM850 delivered the tDCS through electrodes.
- Sham tDCS: Subjects receiving sham transcranial direct current stimulation, had electrodes placed on the subjects head in a manner which caused a temporary "tingling" sensation without effects on the brain. Subjects receiving sham transcranial direct current stimulation underwent 8 sessions during a 2 1/2 week period while "on" medication.
Period: Overall Study
Arm/Group | Real tDCS | Sham tDCS
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Real tDCS: Subjects received real transcranial direct current stimulation
- Sham tDCS: Subjects received sham transcranial direct current stimulation
- Total: Total of all reporting groups
Arm/Group | Real tDCS | Sham tDCS | Total
Number analyzed (Participants) | 13 | 12 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.0) | 64.2 (8.8) | 63.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 7 | 16
Hoehn-Yahr on medication [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided. The measurement on the Hoehn and Yahr was taken while the subject was on medication.
  units on a scale | 2.5 (0.1) | 2.4 (0.2) | 2.42 (0.2)
Hoehn-Yahr off medication [Mean (Standard Deviation); unit: units on scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided. The measurement on the Hoehn and Yahr was taken while the subject was off medication.
  units on scale | 2.7 (0.3) | 2.9 (0.4) | 2.8 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed Before and After Real and Sham tDCS.
Description: Gait speed was measured by the time it took the subject to walk 10m. Subjects were instructed to walk at a fast pace without taking the risk of falling, wearing the same shoes and using assistive devices consistently if needed. Gait speed was measured at baseline and post-tDCS.
Time Frame: baseline, 1 day post, 1 month post, 3 months post-tDCS
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Real tDCS While on Medication: Timed gait during 10m walking task in subjects on medication at baseline, one day post tDCS, one month post tDCS, three month post tDCS.
- Sham tDCS While on Medication: Timed gait during 10m walking task in subjects on medication at baseline, one day post sham tDCS, one month post sham tDCS, three month post sham tDCS.
- Real tDCS While Off Medication: Timed gait during 10m walking task in subjects off medication at baseline, one day post tDCS, one month post tDCS, three month post tDCS.
- Sham tDCS While Off Medication: Timed gait during 10m walking task in subjects off medication at baseline, one day post sham tDCS, one month post sham tDCS, three month post sham tDCS.
Arm/Group | Real tDCS While on Medication | Sham tDCS While on Medication | Real tDCS While Off Medication | Sham tDCS While Off Medication
Number analyzed (Participants) | 13 | 12 | 13 | 12
Seconds
  Baseline | 8.7 (2.4) [-1.6 to 1.6] | 8.6 (2.6) | 9.7 (3.6) | 9.5 (4.1)
  One day post tDCS | 7.2 (1.6) | 7.6 (1.5) | 7.5 (1.5) | 9.8 (4.7)
  One month post tDCS | 7.0 (1.2) | 8.7 (3.7) | 7.6 (1.4) | 10.9 (7.3)
  Three month post tDCS | 7.2 (1.5) | 8.8 (4.2) | 9.0 (4.8) | 9.7 (4.6)

2. Secondary Outcome: UPDRS Total Scores Before and After Real tDCS Course and After Sham tDCS Course.
Description: The Total Unified Parkinson's Disease Rating Scale (UPDRS) is an overall clinical rating scale that quantifies the signs and symptoms of Parkinson's disease. The total UPDRS score was obtained from subject examination, subject interviews and questionnaires. The UPDRS encompasses measurement of mentation, behavior, mood, activities of daily living and motor skills. The total UPDRS scores ranges from 0 (not affected) to 176 (most severely affected). The UPDRS was administred at baseline and at 1 day post, 1 month post, and 3 months post tDCS or sham, while on medication and off medication.
Time Frame: baseline, 1 day post, 1 month post, 3 months post-tDCS
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Real tDCS While on Medication: The total UPDRS score on medication while receiving real tDCS
- Sham tDCS While on Medication: The total UPDRS score on medication while receiving sham tDCS
- Real tDCS While Off Medication: The total UPDRS score off medication while receiving real tDCS
- Sham tDCS While Off Medication: The total UPDRS score off medication while receiving sham tDCS
Arm/Group | Real tDCS While on Medication | Sham tDCS While on Medication | Real tDCS While Off Medication | Sham tDCS While Off Medication
Number analyzed (Participants) | 13 | 12 | 13 | 12
units on a scale
  Baseline | 42.5 (10.8) | 39.5 (12.8) | 58.4 (14.7) | 53.6 (14.5)
  1 day post tDCS | 36.9 (11.1) | 32.0 (11.7) | 54.1 (13.1) | 50.4 (16.2)
  1 month post tDCS | 42.5 (7.8) | 36.1 (11.0) | 56.1 (13.2) | 54.4 (12.1)
  3 months post tDCS | 43.4 (9.1) | 35.5 (13.8) | 60.1 (13.6) | 52.4 (17.0)

3. Secondary Outcome: UPDRS Motor Scores Before and After Real tDCS Course and After Sham tDCS Course.
Description: The Motor Unified Parkinson's Disease Rating Scale (UPDRS) includes only the motor assessment of the UPDRS (Part III) and examines speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability and body bradykinesia. The scores range from 0 (no motor impairment) to 108 (severe motor impairment). The Motor UPDRS was administred at baseline and at 1 day post, 1 month post, and 3 months post tDCS or sham. Subjects were assessed on medication and off medication.
Time Frame: baseline, 1 day post, 1 month post, and 3 months post real and sham tDCS
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Real tDCS While on Medication: The motor UPDRS score on medication while receiving real tDCS
- Sham tDCS While on Medication: The motor UPDRS score on medication while receiving sham tDCS
- Real tDCS While Off Medication: The motor UPDRS score off medication while receiving real tDCS
- Sham tDCS While Off Medication: The motor UPDRS score off medication while receiving sham tDCS
Arm/Group | Real tDCS While on Medication | Sham tDCS While on Medication | Real tDCS While Off Medication | Sham tDCS While Off Medication
Number analyzed (Participants) | 13 | 12 | 13 | 12
units on a scale
  Baseline | 22.2 (8.7) | 17.5 (8.0) | 34.0 (10.0) | 26.5 (8.4)
  1 day post tDCS | 20.4 (7.7) | 15.6 (7.9) | 31.5 (7.3) | 29.0 (11.7)
  1 month post tDCS | 22.7 (6.6) | 18.6 (8.1) | 31.4 (9.9) | 29.0 (8.1)
  3 months post tDCS | 23.1 (7.8) | 17.6 (8.5) | 34.0 (10.3) | 27.1 (10.5)

4. Secondary Outcome: Bradykinesia Measure Before and After Real and Sham tDCS.
Description: Bradykinesia refers to the slowness in executing a movement. Bradykinesia was assessed by measuring the time in seconds it takes to do the following sequence, 10 times: 1) hand closing and opening while squeezing a ball 2) elbow flexion 3) hand closing and opening, and 4) elbow extension. Subjects were allowed to practice these hand and arm movements until performance appeared not to get faster, and then were abstained from further practice to minimize learning effects. The time it takes subjects to execute the entire sequence 10 times with either the left or right arm/hand was measured. Means are reported for each group.
Time Frame: baseline, 1 day post, 1 month post, 3 months post tDCS
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Real tDCS While on Medication: Bradykinesia measured in the hands and arms while on medication and receiving real tDCS.
- Sham tDCS While on Medication: Bradykinesia measured in the hands and arms while on medication and receiving sham tDCS.
- Real tDCS While Off Medication: Bradykinesia measured in the hands and arms while off medication and receiving real tDCS.
- Sham tDCS While Off Medication: Bradykinesia measured in the hands and arms while off medication and receiving sham tDCS.
Arm/Group | Real tDCS While on Medication | Sham tDCS While on Medication | Real tDCS While Off Medication | Sham tDCS While Off Medication
Number analyzed (Participants) | 13 | 12 | 13 | 12
seconds
  Baseline | 12.3 (3.5) | 12.3 (4.0) | 14.5 (4.5) | 14.4 (5.3)
  1 day post tDCS | 8.5 (1.8) | 10.5 (2.3) | 8.9 (1.8) | 11.1 (2.6)
  1 month post tDCS | 9.1 (2.0) | 10.5 (2.3) | 9.4 (1.9) | 11.7 (3.8)
  3 months post tDCS | 9.0 (1.8) | 10.4 (2.5) | 9.7 (2.0) | 11.6 (4.0)

ADVERSE EVENTS:
Arm/Group | Real tDCS | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS (N=13) | Sham tDCS (N=12)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — first degree burn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes